CLINICAL TRIAL: NCT07144553
Title: Examining the Relationship Between Eating Disorders, Anthropometric Characteristics, and Physical Activity After Bariatric Surgery: A 2-Year Longitudinal Study
Brief Title: Relationship Between Eating Disorders, Anthropometric Characteristics, and Physical Activity After Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, İsmail Koç, Assistant Professor, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Other Study IDs: IsmailKoc
Record Dates: First submitted 2025-08-19; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Eating Disorder; Bariatric Surgery
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bariatric Surgery Group: Individuals Undergone Bariatric Surgery

SUMMARY:
In individuals diagnosed with obesity, the traditional treatment method involves changing and regulating dietary habits and increasing physical activity levels. When these measures prove insufficient, pharmacological interventions are used.

When exercise programs conducted after bariatric surgery are compared to weight loss achieved through surgery alone, it is believed that physical activity after bariatric surgery is an effective approach to improving metabolic health.

Gastric leptin level indicates the level of leptin hormone found in stomach tissue. Leptin is a hormone produced by adipose tissue in the body and plays a role in energy balance. It generally controls appetite by reducing feelings of hunger and helps regulate body weight by increasing energy expenditure.

This study aims to examine the relationship between gastric leptin levels, eating disorders, and physical activity after bariatric surgery.

DETAILED DESCRIPTION:
n individuals diagnosed with obesity, the traditional treatment method involves changing and regulating dietary habits and increasing physical activity levels. When these measures prove insufficient, pharmacological interventions are used. However, in 90% of individuals diagnosed with obesity, these treatments have been found to be ineffective, failing to achieve the desired results. It has been reported that weight loss of 5-10% over a five-year period is difficult to achieve. When all these methods are evaluated, it has been reported that bariatric surgery has been a successful technique in improving the health of individuals diagnosed with obesity in recent years. When a technique combining different methods and approaches, such as calorie restriction, physical activity, and behavioral changes in individuals, is attempted, it has been reported that the weight gained in the long term is regained, and the individual is able to perform their physical abilities to a large extent. When exercise programs conducted after bariatric surgery are compared to weight loss achieved through surgery alone, it is believed that physical activity after bariatric surgery is an effective approach to improving metabolic health.

Gastric leptin level indicates the level of leptin hormone found in stomach tissue. Leptin is a hormone produced by adipose tissue in the body and plays a role in energy balance. It generally controls appetite by reducing feelings of hunger and helps regulate body weight by increasing energy expenditure.

This study aims to examine the relationship between gastric leptin levels, eating disorders, and physical activity after bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of obesity and BMI≥ 35 (indication for surgery),
* Indication for bariatric surgery and planned LPSG surgical procedure,
* Age 18 or older,
* Ability to understand and speak Turkish,
* Ability to read and write,

Exclusion Criteria:

* Having undergone orthopedic surgery on the lower extremities,
* Having cardio-respiratory failure that prevents walking,
* Having a musculoskeletal disorder
* Presence of varicose veins,
* Presence of urinary stress incontinence,
* Presence of systemic or rheumatological disease,
* Pregnancy,
* Refusal to participate in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Individuals Undergone Bariatric Surgery
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2025-08-15 (Actual); Primary Completion 2025-08-19 (Actual); Study Completion 2025-08-19 (Actual)

PRIMARY OUTCOMES:
Structural Sociodemographic survey | 2 year
  to get information about physical activity duration and other secondary diseases
Body Mass Index | 2 year
  It will be calculated as weight in kilograms divided by height in meters squared
Eating Disorder Examination Questionnaire | 2 year
  Eating Disorder Examination Questionnaire (EDE-Q). The EDE-Q consists of four subscales: Restraint, Eating Concerns, Weight Concerns, and Shape Concerns. Each item is rated on a 7-point Likert scale ranging from 0 to 6, with higher scores indicating greater severity of eating disorder symptoms. Subscale scores are calculated as the mean of relevant items, and the Global score is the average of the four subscales. Possible range for each subscale and the global score: 0 (no symptoms) to 6 (highest symptom severity).

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Lutfi Kirdar TRH, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No